CLINICAL TRIAL: NCT01178086
Title: Rituximab in the Treatment of Chronic Lymphocytic Leukemia, "CLL NIS"
Brief Title: A Study on Rituximab (MabThera) in Participants With Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22610
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2017-12

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants With CLL: Participants with CLL who are being treated with intravenous (IV) rituximab in combination with chemotherapy, will be observed for 24 months including 6-month treatment period.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab IV
  Other Names: MabThera

SUMMARY:
This observational study will assess the therapeutic efficiency, treatment schedules, handling procedures, and the safety profile of rituximab in routine care in participants with CLL.

ELIGIBILITY:
Inclusion Criteria:

* CLL requiring treatment
* Participants receiving a chemotherapy in combination with rituximab (decision taken by doctor prior to and independent from inclusion in this non-interventional study)
* After this trial started, an amendment to the study protocol was introduced, adding a further inclusion criterion: Comorbidities according to cumulative illness rating scale (CIRS) score greater than (>) 6 and/or creatinine clearance less than (<) 70 milliliters per minute (mL/min)

Exclusion Criteria:

* Participants with contraindication to rituximab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CLL on chemotherapy receiving rituximab
Sampling Method: Probability Sample
Enrollment: 681 (Actual)
Dates: Start 2010-02-22 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PIOH PD Dr. R. Schnell - Dr. H. Schulz - Dr. M. Hellmann, Frechen, Germany

REFERENCES:
- [Derived] Reiser M, Dorfel S, Hensel M, Hoesl M, Jordan WO, Koenigsmann M, Meyer D, Reichert D, Schwarzer A, Marquardt M, Kellershohn K, Jentsch-Ullrich K. Rituximab in combination with chemotherapy for the treatment of chronic lymphocytic leukaemia in clinical practice. Eur J Haematol. 2018 May;100(5):455-464. doi: 10.1111/ejh.13040. Epub 2018 Mar 22. PMID 29393986

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This single arm study had baseline and analysis reported per 2 arms (Unselected Population and "Slow Go" Subpopulation).
Groups:
- Participants With Chonic Lymphatic Leukemia (CLL): Participants with CLL who were treated with intravenous (IV) rituximab in combination with chemotherapy, were observed for 24 months including 6-month treatment period.
Period: Overall Study
Arm/Group | Participants With Chonic Lymphatic Leukemia (CLL)
Started | 681 (Safety analysis set: participants who received at least one dose of rituximab.)
Effectiveness Analysis Set (EAS) | 661 (who received at least 1 dose of rituximab and had data from baseline and at least 1 follow-up visit.)
Completed | 349
Not Completed | 332
Not completed — Participant refusal | 7
Not completed — Physician Decision | 44
Not completed — Switch to other CLL therapy | 113
Not completed — Death | 59
Not completed — Other unspecified | 89
Not completed — Excluded from EAS | 20

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of EAS has been reported.
Groups:
- Unselected Population (Participants With Any Comorbidity): Unselected population (participants with any comorbidity) who were treated with IV rituximab in combination with chemotherapy, were observed for 24 months including 6-month treatment period.
- "Slow Go" Subpopulation: "Slow go" subpopulation (participants with cumulative illness rating scale for geriatrics [CIRS-G] score greater than [>] 6 and/or creatinine clearance less than [<] 70 milliliters per minute [mL/min]) who were treated with IV rituximab in combination with chemotherapy, were observed for 24 months including 6-month treatment period.
- Total: Total of all reporting groups
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation | Total
Number analyzed (Participants) | 472 | 189 | 661
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (9.0) | 74.2 (7.9) | 70.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 84 | 244
  Male | 312 | 105 | 417

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed Using Kaplan-Meier Estimate
Description: PFS was defined as the time from initiation of treatment with rituximab in combination with chemotherapy to disease progression or death due to any cause, whichever occurred first. Disease progression was defined as the occurrence of at least one of the following: greater than or equal to (>/=) 50 percent (%) increase in the longest diameter of at least two enlarged lymph nodes, increase in spleen and/or liver size by at least 2 centimeters (cm) from Baseline as determined by measurement below the costal margin, or >/=50% increase in the number of circulating lymphocytes. Participants without disease progression or death at the time of analysis were censored at the last date of tumor evaluation in terms of PFS.
Time Frame: From initiation of treatment up to disease progression or death due to any cause, whichever occurred first (assessed up to 24 months)
Population: Analysis was performed on EAS.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- "Slow Go" Subpopulation: "Slow go" subpopulation (participants with CIRS-G score >6 and/or creatinine clearance <70 mL/min) who were treated with IV rituximab in combination with chemotherapy, were observed for 24 months including 6-month treatment period.
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 472 | 189
months | 50.6 [42.4 to 59.6] | 33.7 [26.2 to NA] — Data 'not estimable' due to insufficient events since follow-up period was too short.

2. Primary Outcome: Percentage of Participants Without Progression or Death
Description: Disease progression was defined as the occurrence of at least one of the following: >/=50% increase in the longest diameter of at least two enlarged lymph nodes, increase in spleen and/or liver size by at least 2 cm from Baseline as determined by measurement below the costal margin, or >/=50% increase in the number of circulating lymphocytes.
Time Frame: as for outcome 1
Population: Analysis was performed on EAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 472 | 189
percentage of participants | 71.1 [66.1 to 75.5] | 62.7 [53.9 to 70.3]

3. Secondary Outcome: Percentage of Participants With Progression and Death
Description: Percentage of participants with an event (progression or death) was reported. Disease progression was defined as the occurrence of at least one of the following: >/=50% increase in the longest diameter of at least two enlarged lymph nodes, increase in spleen and/or liver size by at least 2 cm from Baseline as determined by measurement below the costal margin, or >/=50% increase in the number of circulating lymphocytes.
Time Frame: as for outcome 1
Population: Analysis was performed on EAS with events.
Measure: Number; unit: percentage of participants
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 106 | 51
percentage of participants
  Progression | 68.9 | 66.7
  Death | 31.1 | 33.3

4. Secondary Outcome: Percentage of Participants Who Received Each Treatment During the Course of Study
Description: The chemotherapeutic regimen administereted during the course of study were: Rituximab-Bendamustine (R-Benda), Rituximab-Fludarabine-Cyclophosphamide (R-FC), Rituximab-Clorambucil (R-Clb), R-Other and Rituximab mono.
Time Frame: Baseline, Cycle 1, 2, 3, 4, 5, 6, 7, 8, last Cycle (Cycle 18) (each cycle=1 month)
Population: Analysis was performed on EAS.
Measure: Number; unit: percentage of participants
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 472 | 189
percentage of participants
  R-Benda at Baseline | 58.5 | 64.0
  R-Benda at Cycle 1 | 56.8 | 60.3
  R-Benda at Cycle 2 | 60.0 | 67.8
  R-Benda at Cycle 3 | 58.8 | 64.8
  R-Benda at Cycle 4 | 57.9 | 62.3
  R-Benda at Cycle 5 | 56.5 | 58.3
  R-Benda at Cycle 6 | 55.3 | 60.6
  R-Benda at Cycle 7 | 44.7 | 29.4
  R-Benda at Cycle 8 | 61.5 | 10.0
  R-Benda at Last Cycle | 55.7 | 62.4
  R-FC at Baseline | 23.3 | 8.5
  R-FC at Cycle 1 | 22.0 | 7.9
  R-FC at Cycle 2 | 24.0 | 9.3
  R-FC at Cycle 3 | 23.5 | 10.9
  R-FC at Cycle 4 | 24.4 | 10.3
  R-FC at Cycle 5 | 23.4 | 10.8
  R-FC at Cycle 6 | 23.4 | 9.2
  R-FC at Cycle 7 | 10.5 | 5.9
  R-FC at Cycle 8 | 3.8 | 0.0
  R-FC at Last Cycle | 23.7 | 8.5
  R-Clb at Baseline | 5.5 | 11.1
  R-Clb at Cycle 1 | 5.5 | 11.1
  R-Clb at Cycle 2 | 5.7 | 9.8
  R-Clb at Cycle 3 | 5.8 | 10.3
  R-Clb at Cycle 4 | 6.4 | 11.0
  R-Clb at Cycle 5 | 6.4 | 11.7
  R-Clb at Cycle 6 | 6.2 | 12.8
  R-Clb at Cycle 7 | 5.3 | 11.8
  R-Clb at Cycle 8 | 7.7 | 20.0
  R-Clb at Last Cycle | 5.5 | 10.6
  R-Other at Baseline | 9.7 | 11.1
  R-Other at Cycle 1 | 9.5 | 9.5
  R-Other at Cycle 2 | 9.3 | 10.9
  R-Other at Cycle 3 | 9.0 | 10.9
  R-Other at Cycle 4 | 8.3 | 10.3
  R-Other at Cycle 5 | 8.8 | 10.8
  R-Other at Cycle 6 | 8.6 | 10.1
  R-Other at Cycle 7 | 10.5 | 5.9
  R-Other at Cycle 8 | 0.0 | 10.0
  R-Other at Last Cycle | 8.9 | 8.5
  Rituximab Mono at Baseline | 0.0 | 0.0
  Rituximab Mono at Cycle 1 | 0.0 | 0.0
  Rituximab Mono at Cycle 2 | 0.7 | 2.2
  Rituximab Mono at Cycle 3 | 2.4 | 3.0
  Rituximab Mono at Cycle 4 | 2.4 | 6.2
  Rituximab Mono at Cycle 5 | 4.6 | 7.5
  Rituximab Mono at Cycle 6 | 6.2 | 7.3
  Rituximab Mono at Cycle 7 | 28.9 | 47.1
  Rituximab Mono at Cycle 8 | 26.9 | 60.0
  Rituximab Mono at Last Cycle | 5.7 | 9.5

5. Secondary Outcome: Mean Body Weight
Time Frame: Baseline, last cycle (Cycle 18) (each cycle=1 month), last visit (follow-up) (24 months)
Population: Analysis was performed on EAS. Overall number of participants analyzed=participants analyzed for this outcome. Here, number analyzed=participants evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 471 | 189
kilograms (kg)
  Baseline | 77.4 (14.1) | 75.0 (14.2)
  Last Cycle: number analyzed (Participants) | 366 | 139
  Last Cycle | 77.4 (15.2) | 73.7 (13.9)
  Last Visit: number analyzed (Participants) | 269 | 99
  Last Visit | 77.0 (15.3) | 73.3 (14.2)

6. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: ECOG performance status was measured on a 4 point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=Capable of only limited self-care, confined to bed/chair >50% of waking hours.
Time Frame: Baseline, last cycle (Cycle 18) (each cycle=1 month), last visit (follow-up) (24 months)
Population: Analysis was performed on EAS. Here, number analyzed=participants evaluable at specified time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 472 | 189
percentage of participants
  Grade 0 at Baseline | 36.4 | 23.8
  Grade 0 at Last Cycle | 23.9 | 19.0
  Grade 0 at Last Visit: number analyzed (Participants) | 371 | 145
  Grade 0 at Last Visit | 34.0 | 26.2
  Grade 1 at Baseline | 40.5 | 45.0
  Grade 1 at Last Cycle | 33.5 | 35.4
  Grade 1 at Last Visit: number analyzed (Participants) | 371 | 145
  Grade 1 at Last Visit | 28.0 | 22.1
  Grade 2 at Baseline | 4.9 | 6.3
  Grade 2 at Last Cycle | 3.4 | 4.8
  Grade 2 at Last Visit: number analyzed (Participants) | 371 | 145
  Grade 2 at Last Visit | 3.8 | 6.9
  Grade 3 at Baseline | 0.4 | 2.1
  Grade 3 at Last Cycle | 1.3 | 1.6
  Grade 3 at Last Visit: number analyzed (Participants) | 371 | 145
  Grade 3 at Last Visit | 1.6 | 2.1
  Missing at Baseline | 17.8 | 22.8
  Missing at Last Cycle | 37.9 | 39.2
  Missing at Last Visit: number analyzed (Participants) | 371 | 145
  Missing at Last Visit | 32.6 | 42.8

7. Secondary Outcome: Percentage of Participants With Karnofsky Performance Status Index
Description: Performance status was reflected by the Karnofsky index. Karnofsky performance status index ranges from 0-100% with higher scores indicating better functional status. An index between 90% and 100% corresponds to ECOG grade 0, index between 70% and 80% corresponds to ECOG grade 1, index between 50% and 60% corresponds to ECOG grade 2, index 40% corresponds to ECOG grade 3. ECOG grade 0=Fully active, able to carry on all pre-disease activities without restriction; grade 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; grade 2=Ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; grade 3=Capable of only limited self-care, confined to bed/chair >50% of waking hours.
Time Frame: Baseline, last cycle (Cycle 18) (each cycle=1 month), last visit (follow-up) (24 months)
Population: Analysis was performed on EAS. Here, number analyzed=participants evaluable at specified time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 472 | 189
percentage of participants
  Karnofsky index 100% at Baseline | 25.4 | 7.4
  Karnofsky index 100% at Last Cycle | 14.8 | 7.9
  Karnofsky index 100% at Last Visit: number analyzed (Participants) | 371 | 145
  Karnofsky index 100% at Last Visit | 17.5 | 11.0
  Karnofsky index 90% at Baseline | 24.4 | 25.4
  Karnofsky index 90% at Last Cycle | 17.4 | 18.5
  Karnofsky index 90% at Last Visit: number analyzed (Participants) | 371 | 145
  Karnofsky index 90% at Last Visit | 14.6 | 11.7
  Karnofsky index 80% at Baseline | 14.2 | 16.9
  Karnofsky index 80% at Last Cycle | 7.4 | 8.5
  Karnofsky index 80% at Last Visit: number analyzed (Participants) | 371 | 145
  Karnofsky index 80% at Last Visit | 7.3 | 9.0
  Karnofsky index 70% at Baseline | 3.4 | 5.8
  Karnofsky index 70% at Last Cycle | 3.0 | 4.2
  Karnofsky index 70% at Last Visit: number analyzed (Participants) | 371 | 145
  Karnofsky index 70% at Last Visit | 2.4 | 2.8
  Karnofsky index 60% at Baseline | 0.6 | 1.1
  Karnofsky index 60% at Last Cycle | 0.2 | 1.6
  Karnofsky index 60% at Last Visit: number analyzed (Participants) | 371 | 145
  Karnofsky index 60% at Last Visit | 0.3 | 0.7
  Karnofsky index 50% at Baseline | 0.2 | 0.0
  Karnofsky index 50% at Last Cycle | 0.2 | 0.0
  Karnofsky index 50% at Last Visit: number analyzed (Participants) | 371 | 145
  Karnofsky index 50% at Last Visit | 0.3 | 0.7
  Karnofsky index 40% at Baseline | 0.0 | 0.0
  Karnofsky index 40% at Last Cycle | 0.0 | 0.0
  Karnofsky index 40% at Last Visit: number analyzed (Participants) | 371 | 145
  Karnofsky index 40% at Last Visit | 0.0 | 0.0
  Missing at Baseline | 31.8 | 43.4
  Missing at Last Cycle | 57.0 | 59.3
  Missing at Last Visit: number analyzed (Participants) | 371 | 145
  Missing at Last Visit | 57.7 | 64.1

8. Secondary Outcome: Percentage of Participants With General Symptoms
Description: General symptoms included fatigue, reduced performance, frequent infections, abdominal pain and exhaustion.
Time Frame: Baseline, last cycle (Cycle 18) (each cycle=1 month), last visit (follow-up) (24 months)
Population: Analysis was performed on EAS. Here, number analyzed=participants evaluable at specified time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 472 | 189
percentage of participants
  Fatigue at Baseline | 38.1 | 45.0
  Fatigue at Last Cycle | 23.5 | 22.8
  Fatigue at Last Visit: number analyzed (Participants) | 371 | 145
  Fatigue at Last Visit | 17.8 | 14.5
  Reduced Performance at Baseline | 46.0 | 49.2
  Reduced Performance at Last Cycle | 24.2 | 20.6
  Reduced Performance at Last Visit: number analyzed (Participants) | 371 | 145
  Reduced Performance at Last Visit | 21.3 | 22.1
  Frequent Infections at Baseline | 13.8 | 15.9
  Frequent Infections at Last Cycle | 5.5 | 4.2
  Frequent Infections at Last Visit: number analyzed (Participants) | 371 | 145
  Frequent Infections at Last Visit | 7.5 | 6.9
  Abdominal Pain at Baseline | 8.3 | 7.9
  Abdominal Pain at Last Cycle | 1.9 | 3.2
  Abdominal Pain at Last Visit: number analyzed (Participants) | 371 | 145
  Abdominal Pain at Last Visit | 4.9 | 2.8
  Exhaustion at Baseline | 35.8 | 40.2
  Exhaustion at Last Cycle | 19.5 | 15.9
  Exhaustion at Last Visit: number analyzed (Participants) | 371 | 145
  Exhaustion at Last Visit | 14.6 | 17.2

9. Secondary Outcome: Percentage of Participants With B-Symptoms
Description: B-symptoms included fever, night sweats, weight loss.
Time Frame: Baseline, last cycle (Cycle 18) (each cycle=1 month), last visit (follow-up) (24 months)
Population: Analysis was performed on EAS. Here, number analyzed=participants evaluable at specified time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 472 | 189
percentage of participants
  Fever at Baseline | 4.0 | 4.8
  Fever at Last Cycle | 3.4 | 2.6
  Fever at Last Visit: number analyzed (Participants) | 371 | 145
  Fever at Last Visit | 2.2 | 0.7
  Night Sweats at Baseline | 29.0 | 25.4
  Night Sweats at Last Cycle | 3.2 | 2.6
  Night Sweats at Last Visit: number analyzed (Participants) | 371 | 145
  Night Sweats at Last Visit | 7.0 | 6.9
  Weight Loss at Baseline | 21.8 | 21.2
  Weight Loss at Last Cycle | 4.2 | 3.7
  Weight Loss at Last Visit: number analyzed (Participants) | 371 | 145
  Weight Loss at Last Visit | 5.7 | 4.1

10. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR)
Description: Response to treatment was assessed as per clinical routine. BOR included complete response(CR or CR with incomplete hematopoietic regeneration),partial response(PR or nodular PR),stable disease(SD),progressive disease(PD). CR:hemoglobin>/=11 grams/deciliter(g/dL), lymphocytes<4000 cells/cubic millimeter(cells/mm^3), neutrophils>5000 cells/mm^3,platelets>100,000 cells/mm^3,bone marrow biopsy with <30% lymphocytes with no lymphocytic infiltrates, no evidence of lymphoid nodules on physical exam, performance status of 0. PR:>50% decrease in size of enlarged lymph nodes, hepatomegaly, splenomegaly, with peripheral counts meeting same criteria as CR or >/=50% improvement from pre-treatment values.PD:occurrence of at least one of following: >/=50% increase in longest diameter of at least 2 enlarged lymph nodes, increase in spleen and liver size by at least 2 cm from Baseline, or >/=50% increase in number of circulating lymphocytes. Participants without CR/PR or PD were considered having SD.
Time Frame: as for outcome 1
Population: Analysis was performed on EAS.
Measure: Number; unit: percentage of participants
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Number analyzed (Participants) | 472 | 189
percentage of participants
  CR | 37.9 | 32.8
  PR | 37.3 | 39.2
  SD | 8.1 | 8.5
  PD | 2.8 | 2.1
  Not assessable | 4.9 | 5.3
  Not assessed / Missing | 9.1 | 12.2

ADVERSE EVENTS:
Time Frame: Baseline up to 24 months
Description: Analysis was performed on safety analysis set.
Arm/Group | Unselected Population (Participants With Any Comorbidity) | "Slow Go" Subpopulation
Serious Adverse Events (participants affected / at risk) | 85/485 | 44/196
Other Adverse Events (participants affected / at risk) | 259/485 | 98/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Unselected Population (Participants With Any Comorbidity) (N=485) | "Slow Go" Subpopulation (N=196)
Anemia (Blood and lymphatic system disorders) | 5 | 6
Autoimmune hemolytic anemia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow toxicity (Blood and lymphatic system disorders) | 1 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 1
Leukopenia (Blood and lymphatic system disorders) | 11 | 5
Neutropenia (Blood and lymphatic system disorders) | 17 | 5
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Adrenal mass (Endocrine disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 1 | 0
Mouth hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 4 | 1
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 2 | 1
Effusion (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 5 | 3
Pyrexia (General disorders) | 13 | 1
Hypersensitivity (Immune system disorders) | 2 | 2
Secondary immunodeficiency (Immune system disorders) | 1 | 1
Atypical Pneumonia (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 10 | 3
Bronchitis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Necrotizing fasciitis (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 3
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Dental operation (Surgical and medical procedures) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Hematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 2
Enterococcal infection (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Hemoglobin decreased (Investigations) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Lymphatic system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalization (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Unselected Population (Participants With Any Comorbidity) (N=485) | "Slow Go" Subpopulation (N=196)
Anemia (Blood and lymphatic system disorders) | 40 | 21
Leukopenia (Blood and lymphatic system disorders) | 129 | 48
Neutropenia (Blood and lymphatic system disorders) | 33 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 99 | 31
Diarrhoea (Gastrointestinal disorders) | 26 | 14
Nausea (Gastrointestinal disorders) | 67 | 20
Chills (General disorders) | 38 | 17
Pyrexia (General disorders) | 46 | 15
Hypersensitivity (Immune system disorders) | 47 | 19
Bacterial infection (Infections and infestations) | 29 | 0
Fatigue (General disorders) | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.